CLINICAL TRIAL: NCT05148221
Title: Mayo Clinic Family Medicine Resident Wellness Study: Feasibility of a Tailored Virtual Exercise Program and Its Impacts on Sleep Patterns and Subjective Mental Fatigue Among Family Medicine Residents: A Step Towards Prevention of Burnout in Early Career Physicians
Brief Title: Mayo Clinic Family Medicine Resident Wellness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Terri Nordin, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-007624
Record Dates: First submitted 2021-10-18; First posted 2021-12-08 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Sleep Patterns
Keywords: Acute and Chronic Cognitive Fatigue; Perceived burnout; Family Medicine Residency Program
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A three-week tailored, virtual exercise intervention. (Experimental): A three-week tailored, virtual exercise intervention.
  Interventions: Other: Questionnaires; Other: Actigraph and activPAL devices

INTERVENTIONS:
Other: Questionnaires — Once each participant signs an informed consent form upon agreeing to participate in the study, they will be asked to complete a simple demographic questionnaire including year in program, work schedule, self-reported height and weight, age, and sex. They will also be interviewed by a faculty of university of Wisconsin-Eau Claire (UWEC) regarding their current and past exercise habits, exercise preferences, and perceived exercise barriers. Two questionnaires listed above (Occupational Fatigue Exhaustion Recovery (OFER 15) and Maslach Burnout Inventory (MBI)) will also be completed by each participant on Qualtrics online platform.
Other: Actigraph and activPAL devices — Actigraph and activPAL devices will be set up based on the demographic information and will be provided to each participant to wear for 7 consecutive days during all waking hours and sleep, except when bathing or swimming. If the first 7-day monitoring period was an overnight inpatient week, the second 7-day monitoring period will be scheduled during a non-overnight week. A day before the first day of the second monitoring period, a new set of Actigraph and activPAL devices will be delivered to each participant. Once the second monitoring period ends, devices will be retrieved from each participant, and data will be downloaded from devices.

SUMMARY:
The objectives of this study are to better understand the association between sleep characteristics (sleep disruptions and deprivations) during overnight shifts and mental fatigue among medical residents, and to explore the feasibility of a virtual, tailored exercise program on sleep characteristics, subjective mental fatigue, and burnout level among residents in family medicine.

DETAILED DESCRIPTION:
The purpose of the proposed study is two-fold: 1) to better understand the association between sleep characteristics (sleep disruptions and deprivations) during overnight shifts and mental fatigue among medical residents; and 2) to explore the feasibility of a three-week tailored, virtual exercise program on sleep characteristics, subjective mental fatigue, and burnout level among residents in family medicine. It is hypothesized that: 1) the greater the number of average sleep disruptions, and the greater the sleep deprivation, the greater the acute mental fatigue during overnight shifts reported by the family medicine residents; 2) the number of average sleep disruptions and the magnitude of sleep deprivation are greater during overnight shifts than non-overnight shifts among family medicine residents; and 3) a three-week tailored virtual exercise program will significantly increase the amount of physical activity throughout the day and reduce the levels of mental fatigue and perceived burnout during overnight shifts.

ELIGIBILITY:
Inclusion Criteria:

• A Family Medicine Resident at the Mayo Clinic Health System of Eau Claire in either the PGY-1 Year, PGY-2 Year, or PGY-2 Year (5 residents from each year).

Exclusion Criteria:

* Participant is not able to wear the devices for the assigned timeframe.
* Any condition the investigator considers will prevent compliance with study instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Work-related mental fatigue | up to 4 weeks
  Subjective work-related mental fatigue will be measured using the OFER 15 which has 15 items on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree). The three subscales of OFER 15 include: chronic fatigue (items 1-5), acute fatigue (items 6-10), and inter-shift recovery (items 11-15) experienced in the past few months. Scores for each subscale range from 0-100. Higher scores indicate acute and chronic fatigue and greater inter-shift recovery.
Work-related burnout | up to 4 weeks
  Levels of burnout will be assessed using the Maslach Burnout Inventory (MBI) which has 22 items on a 7-point Likert scale of 0 (never) to 6 (every day), consisting of three subscales of burnout: emotional exhaustion, depersonalization, and personal accomplishment. Low personal accomplishment scores, high emotional exhaustion scores, and high depersonalization scores suggest increased levels of burnout.

SECONDARY OUTCOMES:
Sleep duration | up to 4 weeks
  Number of hours of sleep per night measured using the activePAL inclinometer
Sleep disruptions | up to 4 weeks
  Number of times shifting from lying to upright posture per night measured using the activePAL inclinometer
Horizontal shifts during sleep per night | up to 4 weeks
  Number of horizontal shifts during sleep per night measured using the active PAL inclinometer

OTHER OUTCOMES:
Exercise duration | up to 4 weeks
  Number of minutes per day of exercise measured by Actigraph wGT3Xbt accelerometer
Exercise Frequency | up to 4 weeks
  Number of days per week of exercise measured by Actigraph wGT3Xbt accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Terri Nordin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System-Eau Claire, Eau Claire, Wisconsin, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials